CLINICAL TRIAL: NCT01944202
Title: Reducing Outpatient Inappropriate Transthoracic Echocardiograms With An Educational Intervention: A Randomized Control Trial
Brief Title: Educational Intervention to Reduce Outpatient Inappropriate Transthoracic Echocardiograms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rory Weiner, MD, Assistant Professor Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2011P001779CR1
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Inappropriate Use of Echocardiography
Keywords: Echocardiography; Appropriate Use Criteria; Educational Intervention
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Intervention (Experimental): Physicians in the intervention arm receive the following multi-faceted educational intervention on transthoracic echocardiogram appropriateness: 1) a lecture at the beginning of the study period, which describes the Appropriate Use Criteria (AUC) for echocardiography and highlights common clinical scenarios for which outpatient TTEs are ordered, 2) an electronic "pocket card" via email that provides tips on appropriate ordering of TTEs, and 3) an individualized monthly feedback report that categorized TTEs ordered over the preceding month. The feedback reports contains the number of TTEs ordered during the month and how many are classified as appropriate, inappropriate, or uncertain based on the 2011 AUC.
  Interventions: Behavioral: Educational intervention
- Control group (No Intervention): Physicians in the control arm have their TTE orders tracked and classified, but do not receive any feedback on their ordering behavior.

INTERVENTIONS:
Behavioral: Educational intervention — Educational and feedback intervention, as described in the Arm Description.
  Arms: Educational Intervention

SUMMARY:
It is well documented that the proportion of inappropriate transthoracic echocardiograms (TTEs) is highest in the ambulatory environment, where it has been reported as high as 30%. Therefore, the potential to improve TTE utilization may be greatest in the outpatient setting. However, no study to date has evaluated whether an Appropriate Use Criteria (AUC)-based educational intervention can reduce inappropriate TTEs in this setting. The investigators therefore designed the first randomized control trial of an AUC-based educational and feedback intervention aimed at reducing inappropriate outpatient TTEs ordered by cardiology and internal medicine physicians in training.

DETAILED DESCRIPTION:
The investigators designed a randomized, control trial of an AUC-based educational and feedback intervention designed to reduce the proportion of inappropriate TTEs in the cardiology and internal medicine outpatient practices at Massachusetts General Hospital. A random number generator divided 24 cardiology fellows and 88 internal medicine residents into control and intervention arms.

During the study, physicians in the intervention arm receive the following multi-faceted educational intervention on TTE appropriateness: 1) a lecture at the beginning of the study period, which describes the AUC for echocardiography and highlights common clinical scenarios for which outpatient TTEs are ordered, 2) an electronic "pocket card" via email that provides tips on appropriate ordering of TTEs, and 3) an individualized monthly feedback report that categorizes TTEs ordered over the preceding month. The feedback reports contain the number of TTEs ordered during the month and how many are classified as appropriate, inappropriate, or uncertain based on the 2011 AUC. A description of all inappropriate TTEs and the rationale for the inappropriate classification is provided. The physicians in the control arm have their TTE orders tracked and classified, but do not receive any feedback on their ordering behavior. While study participants are not blinded to which arm of the study they are in, they were blinded to which arm of the study their colleagues are in.

Prior to the start of the intervention, all study participants receive a knowledge assessment survey. The survey includes five case-based questions designed to assess knowledge of the AUC for TTE and also questions regarding attitudes toward diagnostic testing. Each participant also receives a post-study knowledge assessment survey.

The primary outcome measures in this study are the rate of inappropriate and appropriate TTEs. Secondary outcome measures include the number of TTEs ordered, common appropriate and inappropriate TTE indications, and pre- and post-study knowledge assessment scores among the study physicians.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular Medicine fellows at Massachusetts General Hospital
* Internal Medicine residents at Massachusetts General Hospital

Exclusion Criteria:

* Attending physicians

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate of Inappropriate transthoracic echocardiograms | 9 months
  Rate of inappropriate echocardiograms determined from a review of the electronic medical record.

SECONDARY OUTCOMES:
Rate of Appropriate Transthoracic Echocardiograms | 9 months
  Rate of appropriate transthoracic echocardiograms determined from a review of the electronic medical record.

OTHER OUTCOMES:
Clinical reasons for appropriate and inappropriate transthoracic echocardiograms | 9 months
  All echocardiograms will be classifed according to the Appropriate Use Criteria (AUC). This will allow for determination of the most common clinical indications for both appropriate and inappopriate TTEs.

CONTACTS AND LOCATIONS:
Overall Officials: Rory B Weiner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bhatia RS, Dudzinski DM, Malhotra R, Milford CE, Yoerger Sanborn DM, Picard MH, Weiner RB. Educational intervention to reduce outpatient inappropriate echocardiograms: a randomized control trial. JACC Cardiovasc Imaging. 2014 Sep;7(9):857-66. doi: 10.1016/j.jcmg.2014.04.014. Epub 2014 Aug 13. PMID 25129520